CLINICAL TRIAL: NCT01083810
Title: Evaluation of Kaletra Therapy Over the Long-term
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Dr. Stefan Simianer, Medical Director, Medical Department, Abbott Germany (Wiesbaden)
Other Study IDs: KAL 1 RO; NCT01081470 (obsolete NCT alias); NCT01083836 (obsolete NCT alias)
Record Dates: First submitted 2010-02-26; First posted 2010-03-10 (Estimated); Results first posted 2011-07-29 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; Infection; Kaletra; Resistance; Mutations; alternative Therapy regimen
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections | interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- therapy-naive: Patients who had not received prior antiretroviral drug therapy
  Interventions: Drug: Lopinavir/Ritonavir (Kaletra)
- pre-treated: Patients that had previously received antiretroviral therapy, but are protease inhibitor naive
  Interventions: Drug: Lopinavir/Ritonavir (Kaletra)
- non-B: Patients infected with non-B subtypes of HIV-1
  Interventions: Drug: Lopinavir/Ritonavir (Kaletra)

INTERVENTIONS:
Drug: Lopinavir/Ritonavir (Kaletra) — 3 capsules 2xdaily or 2 tablets 2xdaily Kaletra
  Other Names: ABT-378/r; Kaletra; Lopinavir/Ritonavir

SUMMARY:
Long term observation of patients under lopinavir/ritonavir containing therapy

DETAILED DESCRIPTION:
Three to five year observation of lopinavir/ritonavir therapy. Reporting groups are 1) therapy-naïve patients (144 weeks), 2) therapy-experienced but protease inhibitor naïve patients (240 weeks,) and 3) non-B subtype infected patients (240 weeks).

These three groups of participants with HIV-1 infection were at first registered as three different studies: KAL1RO (this study, NCT01083810, n=137), KAL2RO /KAL5RO (NCT01083836, n=92), and KAL6RO (NCT01081470, n=55) but were now reconciled under KAL1RO (NCT01083810) as a single study with three reporting groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by HIV-1
* Age greater than or equal to 18 years

Exclusion Criteria:

* as described in SmPC (summary of product characteristics) at the time of prescription

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human Immunodeficiency Virus-infected, protease inhibitor-naïve patients from a clinical setting
Sampling Method: Non-Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2001-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Simianer, MD, Study Director — Abbott Germany, Medical Department
Locations (90):
- Germany (90):
  - Site Ref # / Investigator 27706, Aachen
  - Site Ref # / Investigator 52972, Aachen
  - Site Ref # / Investigator 27660, Berlin
  - Site Ref # / Investigator 27937, Berlin
  - Site Ref # / Investigator 52973, Berlin
  - Site Reference ID/Investigator# 27629, Berlin
  - Site Ref # / Investigator 27651, Berlin
  - Site Ref # / Investigator 27912, Berlin
  - Site Reference ID/Investigator# 27544, Berlin
  - Site Reference ID/Investigator# 27567, Berlin
  - Site Ref # / Investigator 27929, Berlin
  - Site Ref # / Investigator 52971, Berlin
  - Site Ref # / Investigator 53468, Berlin
  - Site Ref # / Investigator 27965, Berlin
  - Site Reference ID/Investigator# 27547, Berlin
  - Site Reference ID/Investigator# 27552, Berlin
  - Site Reference ID/Investigator# 27562, Berlin
  - Site Ref # / Investigator 52984, Berlin
  - Site Ref # / Investigator 27639, Berlin
  - Site Ref # / Investigator 52970, Berlin
  - Site Ref # / Investigator 27909, Berlin
  - Site Ref # / Investigator 47113, Berlin
  - Site Reference ID/Investigator# 27574, Chemnitz
  - Site Ref # / Investigator 28060, Cologne
  - Site Ref # / Investigator 52978, Cologne
  - Site Ref # / Investigator 27932, Cologne
  - Site Ref # / Investigator 52979, Cologne
  - Site Ref # / Investigator 48233, Cologne
  - Site Ref # / Investigator 52985, Cologne
  - Site Ref # / Investigator 53464, Cologne
  - Site Ref # / Investigator 27704, Dortmund
  - Site Ref # / Investigator 27947, Dortmund
  - Site Ref # / Investigator 52968, Dortmund
  - Site Reference ID/Investigator# 27558, Duisburg
  - Site Ref # / Investigator 28056, Düsseldorf
  - Site Ref # / Investigator 52983, Frankfurt
  - Site Ref # / Investigator 27928, Frankfurt
  - Site Ref # / Investigator 52967, Frankfurt
  - Site Reference ID/Investigator# 27565, Freiburg im Breisgau
  - Site Reference ID/Investigator# 27566, Fürth
  - Site Ref # / Investigator 53465, Fürth
  - Site Ref # / Investigator 27931, Hamburg
  - Site Ref # / Investigator 27982, Hamburg
  - Site Ref # / Investigator 47114, Hamburg
  - Site Ref # / Investigator 47115, Hamburg
  - Site Reference ID/Investigator# 27551, Hamburg
  - Site Reference ID/Investigator# 27634, Hamburg
  - Site Ref # / Investigator 30864, Hamburg
  - Site Ref # / Investigator 5348, Hamburg
  - Site Reference ID/Investigator# 27546, Hamburg
  - Site Ref # / Investigator 28032, Hamburg
  - Site Ref # / Investigator 52969, Hamburg
  - Site Ref # / Investigator 53467, Hamburg
  - Site Ref # / Investigator 52980, Hamburg
  - Site Ref # / Investigator 27641, Karlsruhe
  - Site Ref # / Investigator 27964, Karlsruhe
  - Site Reference ID/Investigator# 27561, Karlsruhe
  - Site Ref # / Investigator 53466, Koblenz
  - Site Reference ID/Investigator# 27555, Koblenz
  - Site Ref # / Investigator 27905, Krefeld
  - Site Ref # / Investigator 27906, Leipzig
  - Site Ref # / Investigator 52975, Leipzig
  - Site Ref # / Investigator 53463, Leipzig
  - Site Ref # / Investigator 27948, Ludwigshafen
  - Site Ref # / Investigator 52977, Ludwigshafen
  - Site Ref # / Investigator 27902, Mainz
  - Site Reference ID/Investigator# 27543, Mainz
  - Site Ref # / Investigator 28104, Mönchengladbach
  - Site Ref # / Investigator 52981, Mönchengladbach
  - Site Ref # / Investigator 27949, Munich
  - Site Reference ID/Investigator# 27553, Munich
  - Site Ref # / Investigator 27926, Munich
  - Site Ref # / Investigator 53462, Munich
  - Site Ref # / Investigator 27648, Münster
  - Site Reference ID/Investigator# 27568, Münster
  - Site Ref # / Investigator 52982, Nuremberg
  - Site Ref # / Investigator 27988, Oldenburg
  - Site Reference ID/Investigator# 27563, Oldenburg
  - Site Ref # / Investigator 27637, Osnabrück
  - Site Ref # / Investigator 27943, Osnabrück
  - Site Ref # / Investigator 52974, Osnabrück
  - Site Ref # / Investigator 27939, Paderborn
  - Site Ref # / Investigator 27649, Rostock
  - Site Reference ID/Investigator# 27569, Rostock
  - Site Ref # / Investigator 27647, Stuttgart
  - Site Ref # / Investigator 28047, Stuttgart
  - Site Ref # / Investigator 28048, Stuttgart
  - Site Reference ID/Investigator# 27631, Stuttgart
  - Site Ref # / Investigator 52976, Troisdorf
  - Site Ref # / Investigator 27961, Wuppertal

RESULTS

PARTICIPANT FLOW:
Recruitment Details: These three groups of participants with HIV-1 infection were at first registered as three different studies: KAL1RO (this study, NCT01083810, n=137), KAL2RO /KAL5RO (NCT01083836, n=92), and KAL6RO (NCT01081470, n=55) but were now reconciled under KAL1RO (NCT01083810) as a single study with three reporting groups.
Groups:
- Therapy-naive: Participants who had not received prior antiretroviral drug therapy.
- Pre-treated: Participants that had previously received antiretroviral therapy, but were protease inhibitor naive.
- Non-B: Participants infected with non-B subtypes of HIV-1.
Period: Overall Study
Arm/Group | Therapy-naive | Pre-treated | Non-B
Started | 137 | 92 | 55
Completed | 72 | 47 | 35
Not Completed | 65 | 45 | 20
Not completed — Lost to Follow-up | 23 | 11 | 4
Not completed — Adverse Event | 15 | 11 | 4
Not completed — Withdrawal by Subject | 7 | 2 | 4
Not completed — Reason not reported | 6 | 1 | 1
Not completed — Non-compliance | 4 | 7 | 2
Not completed — Simplification | 4 | 1 | 0
Not completed — Death | 2 | 2 | 3
Not completed — Co-morbidities | 1 | 0 | 0
Not completed — Participation in study | 1 | 0 | 0
Not completed — Therapy break | 1 | 2 | 2
Not completed — Virologic failure | 1 | 8 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapy-naive | Pre-treated | Non-B | Total
Number analyzed (Participants) | 137 | 92 | 55 | 284
Age, Customized [Number; unit: Participants]
  >= 18 years of age (exact age not reported) | 137 | 92 | 55 | 284
Sex/Gender, Customized [Number; unit: Participants]
  Female | 17 | 11 | 20 | 48
  Male | 119 | 81 | 35 | 235
  Gender not reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 137 | 92 | 55 | 284

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Virus That Develop Mutations Conferring Resistance to Lopinavir/Ritonavir, NRTIs or NNRTIs
Description: Standard genotypic resistance assays were developed for HIV-1 viral load levels greater than 500 to 1000 copies per milliliter (mL). All 3 protocols recommended this testing be done at Baseline prior to lopinavir/ritonavir therapy and (if possible) in cases of virologic failure. The exact timing varied and depended on whether there was an adequate viral load and physician clinical judgment. Participants with resistance to lopinavir/ritonavir, nucleoside reverse transcriptase inhibitors (NRTI) or non-nucleoside reverse transcriptase inhibitors (NNRTI) at Baseline and follow-up are reported.
Time Frame: Baseline and at any timepoint where testing is possible
Population: All participants with resistance testing at baseline and follow-up are presented.
Measure: Number; unit: Participants
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
Participants
  Genotypic resistance testing performed at Baseline | 137 | 68 | 55
  Complete resistance testing results at Baseline | 122 | 68 | 55
  >Resistance to lopinavir/ritonavir at Baseline | 0 | 2 | 0
  >Partial resistance to NRTI at Baseline | 5 | 0 | 0
  >Partial resistance to NNRTI at Baseline | 0 | 0 | 0
  Underwent resistance testing at follow-up | 2 | 2 | 2
  >Resistance to lopinavir/ritonavir* | 0 | 1 | 0
  >>Resistance to NRTIs | 0 | 1 | 0
  >>Resistance to NNRTIs | 0 | 0 | 0
  *No baseline results avail for this participant | NA — NA=not applicable to this subgroup. | 1 | NA — NA=not applicable to this subgroup.

2. Secondary Outcome: Percentage of Patients With HIV-1 RNA <50 Copies/ml
Description: All 3 protocols recommended that HIV viral load tests be performed at Baseline and each study visit. Study visits were to occur at approximately Weeks 4, 12, and 24, followed by 12-week intervals up to Week 144 in therapy-naive participants and up to Week 240 in the pre-treated and non-B subtype groups. The percentage of participants with HIV-1 ribonucleic acid (RNA) less than 50 copies/mL at each time point is presented by subgroup.
Time Frame: Baseline, Week 4, 12, 24, followed by 12-week intervals up to 144/240 weeks
Population: All participants with HIV-1 RNA measurements at Baseline and any subsequent time point are presented, including those who discontinued due to virologic failure.
Measure: Number; unit: Percentage of participants
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
Percentage of participants
  Baseline | 0 | 3 | 0
  Week 4 | 7 | 26 | 5
  Week 12 | 44 | 38 | 42
  Week 24 | 69 | 58 | 74
  Week 36 | 75 | 60 | 76
  Week 48 | 83 | 67 | 80
  Week 60 | 78 | 65 | 79
  Week 72 | 89 | 62 | 83
  Week 84 | 87 | 66 | 88
  Week 96 | 90 | 58 | 77
  Week 108 | 81 | 66 | 87
  Week 120 | 85 | 63 | 88
  Week 132 | 87 | 52 | 95
  Week 144 | 88 | 65 | 100
  Week 156 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 48 | 100
  Week 168 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 52 | 91
  Week 180 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 53 | 83
  Week 192 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 45 | 100
  Week 204 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 41 | 100
  Week 216 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 50 | 100
  Week 228 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 44 | 75
  Week 240 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 38 | 100

3. Secondary Outcome: Percentage of Patients With HIV-1 RNA 50 to <200 Copies/ml
Description: All 3 protocols recommended that HIV viral load tests be performed at Baseline and each study visit. Study visits were to occur at approximately Weeks 4, 12, and 24, followed by 12-week intervals up to Week 144 in therapy-naive participants and up to Week 240 in the pre-treated and non-B subtype groups. The percentage of participants with HIV-1 RNA levels of 50 to less than 200 copies/mL at each time point is presented by subgroup.
Time Frame: Baseline, Week 4, 12, 24, followed by 12-week intervals up to 144/240 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
Percentage of participants
  Baseline | 1 | 5 | 0
  Week 4 | 17 | 15 | 14
  Week 12 | 32 | 15 | 25
  Week 24 | 22 | 20 | 18
  Week 36 | 18 | 9 | 10
  Week 48 | 10 | 12 | 5
  Week 60 | 13 | 10 | 6
  Week 72 | 5 | 17 | 3
  Week 84 | 9 | 13 | 6
  Week 96 | 6 | 9 | 10
  Week 108 | 14 | 8 | 4
  Week 120 | 5 | 3 | 4
  Week 132 | 3 | 13 | 0
  Week 144 | 0 | 0 | 0
  Week 156 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 0
  Week 168 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 0
  Week 180 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 5 | 8
  Week 192 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 5 | 0
  Week 204 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 6 | 0
  Week 216 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 10 | 0
  Week 228 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 25
  Week 240 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 0

4. Secondary Outcome: Percentage of Patients With HIV-1 RNA 200 to <500 Copies/ml
Description: All 3 protocols recommended that HIV viral load tests be performed at Baseline and each study visit. Study visits were to occur at approximately Weeks 4, 12, and 24, followed by 12-week intervals up to Week 144 in therapy-naive participants and up to Week 240 in the pre-treated and non-B subtype groups. The percentage of participants with HIV-1 RNA levels of 200 to less than 500 copies/mL at each time point is presented by subgroup.
Time Frame: Baseline, Week 4, 12, 24, followed by 12-week intervals up to 144/240 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
Percentage of participants
  Baseline | 0 | 3 | 0
  Week 4 | 18 | 12 | 19
  Week 12 | 12 | 15 | 17
  Week 24 | 3 | 6 | 4
  Week 36 | 1 | 9 | 6
  Week 48 | 1 | 0 | 13
  Week 60 | 2 | 6 | 9
  Week 72 | 0 | 6 | 8
  Week 84 | 2 | 5 | 3
  Week 96 | 0 | 7 | 7
  Week 108 | 0 | 0 | 0
  Week 120 | 2 | 9 | 0
  Week 132 | 3 | 0 | 0
  Week 144 | 0 | 10 | 0
  Week 156 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 10 | 0
  Week 168 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 10 | 0
  Week 180 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 8
  Week 192 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 10 | 0
  Week 204 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 0
  Week 216 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 0 | 0
  Week 228 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 6 | 0
  Week 240 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 6 | 0

5. Secondary Outcome: Percentage of Patients With HIV-1 RNA >500 Copies/ml
Description: All 3 protocols recommended that HIV viral load tests be performed at Baseline and each study visit. Study visits were to occur at approximately Weeks 4, 12, and 24, followed by 12-week intervals up to Week 144 in therapy-naive participants and up to Week 240 in the pre-treated and non-B subtype groups. The percentage of participants with more than 500 HIV-1 RNA copies/mL at each time point is presented by subgroup.
Time Frame: Baseline, Week 4, 12, 24, followed by 12-week intervals up to 144/240 weeks
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
Percentage of participants
  Baseline | 99 | 89 | 100
  Week 4 | 59 | 46 | 63
  Week 12 | 13 | 32 | 15
  Week 24 | 6 | 17 | 4
  Week 36 | 6 | 23 | 8
  Week 48 | 6 | 21 | 3
  Week 60 | 7 | 18 | 6
  Week 72 | 5 | 15 | 6
  Week 84 | 2 | 16 | 3
  Week 96 | 4 | 26 | 7
  Week 108 | 5 | 26 | 9
  Week 120 | 7 | 26 | 8
  Week 132 | 8 | 36 | 5
  Week 144 | 13 | 26 | 0
  Week 156 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 43 | 0
  Week 168 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 38 | 9
  Week 180 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 42 | 0
  Week 192 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 40 | 0
  Week 204 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 53 | 0
  Week 216 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 40 | 0
  Week 228 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 50 | 0
  Week 240 | NA — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 56 | 0

6. Secondary Outcome: Change in Absolute CD4 Cell Count [CD4+ Cells/µL]
Description: The evolution of participants' CD4-positive (CD4+) T-lymphocyte counts after starting the lopinavir/ritonavir-containing regimen was to be assessed by measuring the number of CD4+ cells at baseline and each subsequent study visit. Study visits were to occur at approximately Weeks 4, 12, 24, followed by 12-week intervals up to Week 144 in therapy-naive participants and up to Week 240 in the pre-treated and non-B subtype groups. CD4+ cell count results are reported as the change from Baseline in the absolute number of CD4+ cells per microliter.
Time Frame: Baseline, Week 4, 12, 24, followed by 12-week intervals up to 144/240 weeks
Population: All participants with CD4+ measurements at Baseline and any subsequent time point are included.
Measure: Mean (Standard Deviation); unit: CD4+ cells/µL
Arm/Group | Therapy-naive | Pre-treated | Non-B
Number analyzed (Participants) | 137 | 92 | 55
CD4+ cells/µL
  Baseline | 0 (0) | 0 (0) | 0 (0)
  Week 4 | 140 (145) | 68 (122) | 131 (203)
  Week 12 | 146 (130) | 98 (204) | 92 (117)
  Week 24 | 193 (170) | 106 (209) | 128 (139)
  Week 36 | 211 (203) | 144 (203) | 148 (134)
  Week 48 | 240 (162) | 114 (200) | 204 (173)
  Week 60 | 266 (185) | 144 (196) | 222 (206)
  Week 72 | 248 (201) | 179 (193) | 259 (204)
  Week 84 | 295 (248) | 181 (176) | 226 (161)
  Week 96 | 296 (190) | 192 (223) | 239 (205)
  Week 108 | 329 (204) | 223 (227) | 255 (195)
  Week 120 | 316 (177) | 217 (206) | 275 (199)
  Week 132 | 313 (237) | 213 (167) | 325 (218)
  Week 144 | 292 (163) | 251 (244) | 320 (131)
  Week 156 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 220 (183) | 404 (162)
  Week 168 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 190 (156) | 426 (189)
  Week 180 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 174 (225) | 422 (135)
  Week 192 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 192 (186) | 474 (162)
  Week 204 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 131 (244) | 420 (172)
  Week 216 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 210 (243) | 395 (230)
  Week 228 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 208 (345) | 399 (93)
  Week 240 | NA (NA) — Values not available (NA) as data were collected out to Week 144 in the subgroup of therapy-naive participants. | 179 (185) | 542 (188)

ADVERSE EVENTS:
Time Frame: Investigators were instructed to report adverse events throughout the study (up to 5 years).
Description: Three studies in different populations of participants with HIV-1 infection were conducted in parallel: KAL1RO (NCT01083810, n=137), KAL2RO /KAL5RO (NCT01083836, n=92), and KAL6RO (NCT01081470, n=55). Safety data were collected in a manner that prevented separate analyses for each study, therefore pooled safety data (n=284) are shown.
Groups:
- HIV-infected Patients: Participants with HIV-1 infection, pooled from 3 studies in different populations conducted in parallel: KAL1RO (therapy-naive, NCT01083810, n=137), KAL2RO /KAL5RO (pre-treated, NCT01083836, n=92), and KAL6RO (non-B subtype, NCT01081470, n=55).
Arm/Group | HIV-infected Patients
Serious Adverse Events (participants affected / at risk) | 16/284
Other Adverse Events (participants affected / at risk) | 56/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-infected Patients (N=284)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Ataxia left leg (Nervous system disorders) | 1 (1)
Paralysis left upper extremity (Nervous system disorders) | 1 (1)
Paralysis of left side of face (Nervous system disorders) | 1 (1)
Fall (Nervous system disorders) | 1 (1)
Stupor (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Thickening of meninges (Nervous system disorders) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Lymph nodes enlarged (Blood and lymphatic system disorders) | 1 (1)
Common cold (Infections and infestations) | 1 (1)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1)
Myobacterium avium (Infections and infestations) | 3 (3)
Myobacterium kansaii (Infections and infestations) | 1 (1)
Pneumocystis pneumonia (Infections and infestations) | 4 (5)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Tuberculosis (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1)
Polyserositis (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbosacral syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Cholestasis (Hepatobiliary disorders) | 1 (1)
Gallstones (Hepatobiliary disorders) | 1 (1)
Liver damage (Hepatobiliary disorders) | 1 (1)
Icterus (Hepatobiliary disorders) | 1 (1)
Deep venous thrombosis femoral (Vascular disorders) | 1 (1)
Pulmonary artery thrombosis (Vascular disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Peripheral edema (General disorders) | 1 (1)
Somnolence (General disorders) | 2 (2)
Night sweats (General disorders) | 2 (2)
Reduced general condition (General disorders) | 1 (1)
Shivering (General disorders) | 1 (1)
Fever (General disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV-infected Patients (N=284)
Diarrhea (Gastrointestinal disorders) | 40 (42)
Nausea (Gastrointestinal disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.